CLINICAL TRIAL: NCT06155500
Title: Long-term Follow-up (LTFU) of Patients Treated With Genome-edited Autologous Hematopoietic Stem and Progenitor Cells (HSPC)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CADPT03A12001
Record Dates: First submitted 2023-11-24; First posted 2023-12-04 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Sickle Cell Disease
Keywords: Gene therapy; genome-edited hematopoietic stem and progenitor cellular therapy; sickle cell; autologous transplant; BCL11A
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- OTQ923 (Experimental): Patients were administered OTQ923 while enrolled on the treatment protocol (CADPT03A12101). Patients enrolled on this LTFU study will not be administered any study treatment.
  Interventions: Biological: OTQ923

INTERVENTIONS:
Biological: OTQ923 — There is no treatment allocation. Patients administered were OTQ923 while enrolled on the treatment protocol CADPT03A12101 (NCT04443907)

SUMMARY:
CADPT03A12001 is a prospective, multi-center study that is designed to follow all enrolled patients who have received treatment with OTQ923 for long-term safety and efficacy.

DETAILED DESCRIPTION:
This study is monitoring patients treated with OTQ923, an investigational drug product of ex vivo genome-edited autologous hematopoietic stem and progenitor cells (HSPCs) that induces fetal hemoglobin (HbF) production, for a total of 15 years following infusion to monitor long-term safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have received gene therapy treatment from the parent treatment protocol (CADPT03A12101).
2. Patients must provide informed consent prior to their entry into this study.

Exclusion Criteria:

1. Completion of less than 1 year of safety follow-up in the treatment protocol (CADPT03A12101).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2024-04-16 (Actual); Primary Completion 2039-01-11 (Estimated); Study Completion 2039-01-11 (Estimated)

PRIMARY OUTCOMES:
Number of participants with delayed adverse events that are suspected to be related to previous OTQ923 therapy | Up to 15 years
  Number of participants with delayed adverse events including new secondary malignancies, new incidence or exacerbation of a prior autoimmune disorder, new incidence or exacerbation of a prior rheumatologic disorder, new hematologic disorder, and other adverse events considered to be related to OTQ923 therapy.

SECONDARY OUTCOMES:
Persistence of fetal hemoglobin expression | Up to 15 years
  Assessment of fetal hemoglobin (HbF) expression persistence in peripheral blood will be done by assessing hemoglobin fractionation
WBC chimerism in peripheral blood | 5 years
  Concern for loss of engraftment by monitoring the WBC chimerism annually. Modified white blood cells (WBCs) measured by droplet digital PCR (ddPCR) and NGS will be performed annually through year 5 with subsequent samples stored and run annually in the event of concern for loss of engraftment

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (3):
- United States (3):
  - University of Chicago, Chicago, Illinois
  - Memorial Sloan Kettering Cancer Ctr, New York, New York
  - St Jude Childrens Research Hospital, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No